CLINICAL TRIAL: NCT06142552
Title: Multicenter Study to Evaluate the Efficacy, Safety, Immunogenicity, and Pharmacokinetics of Recombinant Human Coagulation Factor Ⅷ-Fc Fusion Protein (FRSW117) for Injection in Patients With Severe Hemophilia A (Adults and Adolescents)
Brief Title: Phase 3 Clinical Project of Pegylated Recombinant Human Coagulation Factor VIII-Fc Fusion Protein
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS-117-III01
Record Dates: First submitted 2023-11-07; First posted 2023-11-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Severe Hemophilia A
Keywords: Pharmacokinetics; Safety; immunogenicity; effectiveness
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prevention and Treatment Group (PPX group) (Experimental): Subjects received single and multiple doses of 50 IU/kg FRSW117 at first administration of V1 (D1), V4 (18w), and V7 (50w), and PK samples were collected until 168 h post-administration, respectively.
  During prophylaxis, FRSW117 is used for breakthrough therapy if the subject has a breakthrough bleeding event (i.e., a bleeding event during prophylaxis) that requires treatment.
  Interventions: Drug: FRSW117
- On Demand/Preventive Treatment Group (On Demand /PPX Group) (Experimental): The appropriate dose and frequency of administration of FRSW117 is recommended until bleeding events are controlled or returned to pre-bleeding activity.
  Interventions: Drug: FRSW117
- Perioperative management (Experimental): Patients in the PPX and on demand /PPX groups will be allowed to undergo surgery (both major and minor) during the main trial period (prior to 50w), while FRSW117 will be administered perioperatively
  Interventions: Drug: FRSW117

INTERVENTIONS:
Drug: FRSW117 — once a week, 50 weeks and as needed
  Other Names: Recombinant human coagulation factor Ⅷ-Fc fusion protein for injection

SUMMARY:
To evaluate the prophylactic efficacy of recombinant human coagulation factor Ⅷ-Fc fusion protein (FRSW117) for injection in patients with severe hemophilia A.

To evaluate the safety of recombinant human coagulation factor Ⅷ-Fc fusion protein (FRSW117) for injection in patients with severe hemophilia A.

Secondary purpose:

To evaluate the efficacy of recombinant human coagulation factor Ⅷ-Fc fusion protein for injection (FRSW117) in hemostasis and surgical hemostasis in patients with severe hemophilia A.

To evaluate the pharmacokinetic (PK) characteristics of recombinant human coagulation factor Ⅷ-Fc fusion protein (FRSW117) for injection in treated patients with severe hemophilia A.

To evaluate the immunogenicity of recombinant human coagulation factor Ⅷ-Fc fusion protein (FRSW117) for injection in treated patients with severe hemophilia A.

ELIGIBILITY:
inclusion Criteria：

* 12≤ age ≤65 year-old men;
* Patients with clinically confirmed severe hemophilia A, i.e. at screening (central laboratory testing) or previous medical records confirm: FⅧ activity < 1%；
* Previous documented treatment with any recombinant and/or blood-derived coagulation factor Ⅷ products or cryoprecipitation products and dosed ≥150 exposure days (EDs≥150)
* Normal prothrombin time (PT) or International Normalized Ratio (INR)<1.3
* Bleeding events were recorded in detail for at least 6 months prior to screening（Participants in the on demand /PPX group were required to have at least 6 episodes of spontaneous bleeding within 6 months）
* Fully understand and know about this study and sign informed consent to participate in the clinical study voluntarily, subject and/or their guardian can cooperate with them for bleeding treatment at home, and have the ability to complete all study procedures

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug or its excipients, including mouse or hamster proteins;
2. Hypersensitivity or anaphylaxis after FⅧ or IgG2 injection in the past;
3. FⅧ inhibitor positive (≥0.6 BU/mL) during the screening period, or have a history of FⅧ inhibitor positive in the past, or a family history of FⅧ inhibitor positive;
4. Von Willebrand factor (vWF) antigen test results were lower than the lower limit of normal value;
5. Severe anemia at the screening stage (hemoglobin < 60 g/L);
6. Platelet count during screening period < 100×109 /L;
7. Abnormal liver function:

   .Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) >3 times upper limit of normal (ULN); or Serum total bilirubin (TBIL) >1.5x ULN;
8. Patients with abnormal renal function:

   Creatinine clearance (Ccr) <50 ml/min (according to Cockcroft and Gault formula); orSerum creatinine (Cr) >1.5x ULN;
9. People with active hepatitis C, that is, hepatitis C virus (HCV) antibody positive and HCV RNA positive; Or anti-treponema pallidum specific antibody (TPHA) positive; Or positive for antibodies against the human immunodeficiency virus (HIV);
10. Patients with coagulation dysfunction other than hemophilia A;
11. Have a medical condition that may increase the risk of bleeding;
12. A history of drug or alcohol abuse;
13. Have a known mental disorder that may affect trial compliance;
14. Patients who have received transfusions of blood or blood components within 4 weeks prior to screening;
15. Participants who had participated in other clinical trials within 1 month before screening;
16. Use of any anticoagulant or antiplatelet drugs, off-label maximum dose of non-steroidal anti-inflammatory drugs (NSAID) within 7 days prior to screening; Or patients who need to be treated with anticoagulant or antiplatelet drugs or off-label maximum doses of SAID during clinical trials;
17. Severe cardiovascular and cerebrovascular disease or major thromboembolic events, such as stroke, myocardial infarction, unstable angina, congestive heart failure (New York Heart Association [NYHA] grade ≥ III), and severe arrhythmias (including QTc interphase > 480 ms, corrected by Fridericia formula), uncontrolled hypertension (systolic ≥ 160 mmHg or diastolic ≥100 mmHg), deep vein thrombosis, etc.
18. Study patients who had used emesezumab within 6 months prior to first administration of the drug;
19. Patients who had used monoclonal antibody therapy, Fc fusion protein products (except FRSW107 and FRSW117), PEG products (except FRSW117), or intravenous immunoglobulin infusion within 3 months before the first administration of the investigational drug;
20. Study patients who underwent major surgery within 3 months prior to initial drug administration (major surgery is defined in 6.2.3 Perioperative management);
21. Study patients who have used FⅧ preparation of any standard half-life (e.g., Bycoch, Coproch, Biinidin, Renjie, NoL, Antaine, etc.) within 3 days or 5 half-lives prior to first administration of the drug (taking the elderly); Patients who have used any other extended half-life preparation FⅧ within 4 days or 5 half-lives prior to first dosing (for the elderly);
22. Study patients with fever, severe active bacterial or viral infection, and allergies within 2 weeks before the first administration of the drug;
23. Systemic immunomodulators (such as glucocorticoids [> 10 mg/ day equivalent dose of prednisone], alpha-interferon, immunoglobulin, cyclophosphamide, cyclosporin, etc.) used within 14 days prior to the first administration of the study drug or planned during the study period were allowed to be inhaled, nasal spray, or topical corticosteroids;
24. Those who had been vaccinated within 4 weeks prior to initial administration of the study drug; Or who plan to be vaccinated during PK blood collection (only for subjects in the PK subgroup);
25. Plan to have a child or sperm donation during the entire trial period and within 3 months after the last dose, or do not want to use effective physical contraception (such as condoms, diaphragms, Iuds, etc.);
26. Have other serious medical conditions that the researchers said could not benefit from them
27. Subjects deemed unsuitable by other investigators.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
ABR | 1year
  Annual rate of bleeding (ABR) during preventive treatment = Number of bleeding during the efficacy evaluation period/(number of treatment days /365.25)
Effective rate of bleeding treatment | 2year
  The hemostatic effect was evaluated according to a four-level scoring scale, including breakthrough bleeding treatment during preventive treatment and on-demand treatment during on-demand treatment
Safety evaluation | 3year
  Incidence of positive FⅧ inhibitor.
  Adverse events/Adverse events: Adverse events during treatment (TEAE), serious Adverse events (SAEs), adverse events of particular concern (AESI), occurrences of adverse events that cause subjects to discontinue medication, drop out of the study, and death, and occurrences of the above metrics associated with the investigational drug.
  Injection site reaction.
  Laboratory tests: blood routine, urine routine, blood biochemistry, coagulation function, virology and immune function tests.
  Thrombosis markers.
  Vital signs, physical examination, neurological examination, 12-lead electrocardiogram, surgery-related complications.
  PEG level.
Adverse events/reactions | ALL
  Adverse events during treatment (TEAE), serious Adverse events (SAEs), with a special focus on adverse events (AESI), adverse events that cause subjects to discontinue medication, drop out of the study, and die, etc.
Immunogenicity evaluation | ALL
  The positive rate of anti-FRSW117 antibody, anti-PEG antibody and anti-CHO antibody; When the anti-FRSW117 antibody was positive, the anti-RHFVIII antibody and anti-PEG antibody were further detected to evaluate the positive incidence

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Study Chair — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College.
Locations (28):
- China (28):
  - Beijing tongren hospital,CMU, Beijing
  - XiangYa Hospital CentralSouth University, Changsha
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Jinan central hospital, Jinan
  - The First Affiliated Hospital of Shandong First Medical University, Jinan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - The First Hospital of Lanzhou University, Lanzhou
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai
  - Shenzhen Second People's Hospital, Shenzhen
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The Second Hospital of Shanxi Medical University, Taiyuan
  - North China University of Science and Technology Affiliated Hospital, Tangshan
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin
  - Affiliated Hospital of Jiangnan University, Wuxi
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhenyu Li, Xuzhou
  - Subei People's Hospital of Jiangsu province, Yangzhou
  - Henan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhengzhou People's Hospital, Zhengzhou